CLINICAL TRIAL: NCT04470596
Title: Clinical Evaluation of Early Onset Neonatal Infection
Acronym: CLEEONI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CLEEONI
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early bacterial neonatal infection (INBP) defined as occurring in the first 3 days and by extension in the first week of life, remains to this day the leading cause of neonatal morbidity and mortality in developed countries. The germs most frequently found are Streptococcus B (SB) for term newborns (> 37 Weeks of Amenorrhea SA) and Escherichia coli (E. coli) in premature newborns. Although in France, its incidence of 0.4 / 1000 is lower than in other developed countries (0.8 / 1000 general incidence), it remains a major public health concern.

The infection criteria were defined by the National Agency for Health Accreditation and Assessment (ANAES) in 2002, allowing to differentiate between proven infections and highly probable cases of infection. Infection is considered to be proven when SB or E. coli is detected in blood culture or in cerebrospinal fluid. An infection is considered to be highly probable in the event of association of clinical signs (fever, polypnea, desaturation, tachycardia, etc.) evoking a beginning sepsis associating with a disturbance of the biological balance sheet (elevation of CRP, hyperleukocytosis, evidence of colonization on peripheral samples). These criteria remain valid to this day to define the infection.

In order to define the newborns to be monitored, risk factors were established after a review of the literature in 2002. They make it possible to decide on diagnostic management and / or the setting up of a treatment.

Since the recommendations of the ANAES of 2002, the rule, from the presence of a major criterion, was to carry out bacteriological samples peripheral to the birth (gastric liquid, swab of ear and anus) and to systematically collect a CRP of the child between H12 and H48. In the presence of an isolated minor risk factor, simple clinical monitoring (routine) was recommended for 48 hours without deciding firmly on the need for a biological sample. However, it is important to note that these two categories of signs are defined and classified in descending order of risk. This classification does not prejudge a systematic therapeutic attitude. In many situations, the choice is actually left to the practitioner depending on the context.

In 2017, new recommendations were implemented by the French Society of Pediatrics (SFP) and the French Society of Neonatology (SFN) regarding the prevention of INBP. These take up the risk factors of the 2002 ANAES by adding PCR SB at the same level as the traditional PV. They define 3 categories of children according to the risk of INBP and the associated care.

In most cases, these new practices make it possible to dispense with costly blood and bacteriological samples, which cause discomfort and pain for children. In addition, the use of gastric fluid is not internationally validated, its use in the management case remains very controversial. In case of delayed CRP or positive peripheral samples to the germs generated, and even in the absence of clinical signs, antibiotic therapy was almost systematically initiated. Unnecessary exposure to antibiotics promotes the development of bacteriological resistance and unbalances the neonatal flora.

Following the implementation of these new recommendations at the Notre Dame de Bon Secours maternity hospital, which is the case in few centers today and no national survey has yet been carried out on their application, it therefore seems necessary to us evaluate the application of these new recommendations and verify that they allow the detection of all probable or proven infections.

ELIGIBILITY:
Inclusion Criteria:

* Newborns over 36 weeks old, born between 01/01/2019 and 31/12/2019 at the GHPSJ maternity
* Newborn having benefited from close infectious surveillance according to the criteria of the 2017 recommendations (Groups B and C)
* In birth suites near their mother
* Francophone parents

Exclusion Criteria:

* Parents objecting to participation in the study
* Parents deprived of their liberty
* Parents under guardianship or curatorship

Min Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Newborns over 36 weeks old, born between 01/01/2019 and 31/12/2019 at the GHPSJ maternity, having benefited from close infectious surveillance according to the criteria of the 2017 recommendations (Groups B and C).
Sampling Method: Non-Probability Sample
Enrollment: 936 (Actual)
Dates: Start 2020-08-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Newborn screening | Month 3
  This outcome corresponds to percentage of asymptomatic infants at risk for INBP in whom close clinical surveillance has shown no signs of infectious disease, and who have had a probable or proven infection between the discharge from maternity and the age of 1 and 3 months.

SECONDARY OUTCOMES:
negative predictive value of SB PCR for children with proven group B Streptococcus infection | Month 3
  This outcome corresponds to percentage of newborns infected with group B Streptococcus (proven infection) during the postnatal stay and whose mothers' PCRs were negative per partum, whether or not they were monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth WALTER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Weston EJ, Pondo T, Lewis MM, Martell-Cleary P, Morin C, Jewell B, Daily P, Apostol M, Petit S, Farley M, Lynfield R, Reingold A, Hansen NI, Stoll BJ, Shane AL, Zell E, Schrag SJ. The burden of invasive early-onset neonatal sepsis in the United States, 2005-2008. Pediatr Infect Dis J. 2011 Nov;30(11):937-41. doi: 10.1097/INF.0b013e318223bad2. PMID 21654548
- [Result] Stoll BJ, Hansen NI, Sanchez PJ, Faix RG, Poindexter BB, Van Meurs KP, Bizzarro MJ, Goldberg RN, Frantz ID 3rd, Hale EC, Shankaran S, Kennedy K, Carlo WA, Watterberg KL, Bell EF, Walsh MC, Schibler K, Laptook AR, Shane AL, Schrag SJ, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Early onset neonatal sepsis: the burden of group B Streptococcal and E. coli disease continues. Pediatrics. 2011 May;127(5):817-26. doi: 10.1542/peds.2010-2217. Epub 2011 Apr 25. PMID 21518717
- [Result] El Helali N, Nguyen JC, Ly A, Giovangrandi Y, Trinquart L. Diagnostic accuracy of a rapid real-time polymerase chain reaction assay for universal intrapartum group B streptococcus screening. Clin Infect Dis. 2009 Aug 1;49(3):417-23. doi: 10.1086/600303. PMID 19580414